CLINICAL TRIAL: NCT01020968
Title: Catheter-based Transendocardial Delivery of Autologous Bone Marrow-Derived Cells in Patients With Heart Failure Due to Dilated Cardiomyopathy
Brief Title: Use of Ixmyelocel-T (Formerly Catheter-based Cardiac Repair Cell [CRC]) Treatment in Patients With Heart Failure Due to Dilated Cardiomyopathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vericel Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABI-55-0811-1
Record Dates: First submitted 2009-11-25; First posted 2009-11-26 (Estimated); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Dilated Cardiomyopathy
Keywords: Ischemic Dilated Cardiomyopathy; Non-Ischemic Dilated Cardiomyopathy; ixmyelocel-T
MeSH Terms: conditions — Cardiomyopathy, Dilated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ixmyelocel-T (Experimental): The treatment arm of the study will receive catheter-based injections of the study cellular product.
  Interventions: Biological: Ixmyelocel-T
- Vehicle Control (Placebo Comparator): will receive approximately 12-20 intramyocardial injections of 0.4 mL each of vehicle control.
  Interventions: Other: Vehicle Control

INTERVENTIONS:
Biological: Ixmyelocel-T — CRCs will be administered via catheter-based injection to the endocardial surface of the left ventricle.
  Arms: Ixmyelocel-T
Other: Vehicle Control — will receive approximately 12-20 intramyocardial injections of 0.4 mL each of vehicle control into the left ventricle.
  Arms: Vehicle Control

SUMMARY:
This study is designed to assess the safety profile and the efficacy of cardiac repair cells (CRCs) administered via catheter in treating patients with dilated cardiomyopathy (DCM).

DETAILED DESCRIPTION:
Heart failure remains a major public health problem, affecting 5 million patients in the US, with 550,000 new diagnoses made each year (Hunt SA; et al., 2005). Heart failure is the leading cause of hospitalization in persons over 65 years of age with cost exceeding $29 billion annually. Prognosis is very poor once a patient has been hospitalized with heart failure. The mortality risk after heart failure hospitalization is 11.3% at 30 days, 33.1% at 1 year and well over 50% within 5 years (Hunt SA; et al., 2005). These numbers emphasize the need to develop and implement more effective treatments to manage heart failure.

Aastrom is targeting a subset of heart failure patient population, namely those diagnosed with dilated cardiomyopathy. The World Health Organization (WHO) defines dilated cardiomyopathy (DCM) as a cardiac condition wherein a ventricular chamber exhibits increased diastolic and systolic volume and a low (<40%) ejection fraction (Manolio TA; et al., 1992; Towbin JA; et al., 2006). DCM is reported to affect 108,000 to 150,000 patients in the United States (Richardson P; et al., 1996; Towbin JA; et al., 2006).

This study is a prospective, stratified, randomized, open-label, controlled, multi-center study to assess the safety profile and the efficacy of CRCs administered via catheter in treating patients with DCM. Two strata will be used: ischemic (IDCM) and non-ischemic (NIDCM). Within each stratum, patients will be randomized to receive either CRC treatment or control in a 2:1 ratio (8 patients per CRC treatment group and 4 patients per control group). It will enroll a total of 24 patients at 2 sites in the U.S.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ischemic or non-ischemic dilated cardiomyopathy according to WHO criteria. Ischemic: DCM in a patient with a history of myocardial infarction or evidence of clinically significant (>/= 70% narrowing of a major epicardial artery) coronary artery disease. Non-ischemic: Dilation and impaired contraction of left ventricle or both ventricles of idiopathic, familial/genetic, viral and/or immune, toxic origin, or associated with recognized cardiovascular disease in which the degree of myocardial dysfunction is not explained by normal loading conditions or the extent of ischemic damage.
* No other cardiac surgery or percutaneous cardiac interventions likely to produce clinical improvement, as determined by an interventional cardiologist (for PTCA) and a cardiothoracic surgeon (for CABG). This condition is satisfied in patients w/chronic ischemic disease who have previously been successfully revascularized but have failed to show clinical improvement. All patients who are candidates for revascularization are ineligible for participation.
* LVEF </= 30% by echocardiogram within 30 days prior to randomization.
* Symptomatic heart failure in NYHA class III or IV.
* Able to comply with scheduled visits in cardiac out-patient clinic.
* Able to tolerate study procedures, including bone marrow aspiration, cardiac CT, metabolic stress test,6 minute walk test.
* Males and females, 18-86 years of age.
* Life expectancy of 6 months or more in the opinion of the investigator.
* Able to give informed consent.
* Normal organ and marrow function (Leukocytes >/= 3,000/microgram, Absolute neutrophil count >/= 1,500/microgram, Platelets >/= 140,000/microgram, AST(SGOT)/ALT (SGPT) </= 2.5 X institutional standards range and Creatinine </= 2.5 mg/dL).
* Controlled blood pressure (systolic blood pressure </= 140; diastolic blood pressure </= 90 mmHg) and established anti-hypertensive therapy as necessary prior to entry into the study.
* Stable, standard medical therapy for DCM for at least 1 month with NO new medications to treat the disease introduced in the last 3 months. Standard medical therapy includes: Placement of AICD unless contraindicated (refusal of AICD not considered valid contraindication), use of ACE inhibitors and/or AT-1 receptor blockers as well as loop diuretics unless contraindicated and, depending on the type of heart failure associated with the disease, standard therapy may also include use of vasodilators, beta blockers, digoxin, and aldosterone or other medications.
* Pre-existing conditions are adequately controlled in the opinion of the investigator.
* Fertile patients must agree to use an appropriate form of contraception while participating in the study.

Exclusion Criteria:

* Severe primary valvular heart disease including, but not limited to, aortic valve stenosis and insufficiency.
* Known history of COPD defined as Gold stage IIB (FEV1/FVC<70% with 30%</=FEV1<50% predicted, with or without chronic symptoms of cough, sputum production, dyspnea) or more severe or restrictive pulmonary disease.
* Known history of primary pulmonary hypertension.
* VAD implantation.
* Myocardial infarction within 4 weeks prior to randomization.
* History of life-threatening ventricular arrhythmia, except if an AICD is implanted.
* Unstable angina, characterized by increasingly frequent episodes with modest exertion or at rest, worsening severity, and prolonged duration.
* Patients at high risk for complications due to injection procedure (e.g. patients who have severe peripheral atherosclerotic disease that does not allow advancement of the catheter; patients who have a prosthetic aortic or mitral valve; patients who have a LV thrombus or aneurysm; patients who have an aortic dissection or aneurysm, etc.).
* Patients w/poorly controlled diabetes mellitus (HbAlc>9.0%).
* Patients receiving treatment with hematopoietic growth factors (e.g. EPO, G-CSF).
* Patients who require uninterruptible anticoagulation therapy (e.g. warfarin)that cannot be stopped for 72 hours prior to bone marrow aspiration and intramyocardial injections; OR patients receiving anti-platelet therapy (e.g. clopidogrel) that cannot be stopped for 7 days prior to bone marrow aspiration and transendocardial injections, unless contraindicated.
* Known cancer and undergoing treatment including chemotherapy and radiation.
* Patients requiring continuous, systemic, high dose corticosteroid therapy (more than 7.5 mg/day) within 1 month before aspiration or 6 months after injection procedure.
* End stage renal disease requiring dialysis.
* Patients pregnant or lactating; positive for hCG
* History of alcohol consumption regularly exceeding the equivalent of 2 drinks/day (1 drink = 5 oz of wine or 12 oz [360mL] of beer or 1.5 oz [45mL]) of hard liquor or history of illicit drug use w/in 6 months of screening.
* Known allergies to protein products (horse or bovine serum, or porcine trypsin) used in the ex-vivo cell production process.
* BMI of 40 Kg/m2 or greater.
* Patients receiving experimental medications or participating in another clinical study within 30 days of screening.
* HIV or syphilis, positive at time of screening.
* Active Hepatitis B or Hepatitis C infection at the time of screening.
* Patient determined unsuitable for cellular therapy, in the opinion of the investigator or sponsor.
* Patients receiving anti-angiogenic drugs (e.g. anti-VEGF).
* Known allergy or sensitivity to contrast agents used in imaging procedures.
* Minimum LV wall thickness of less than 6mm as determined by ECHO.

Ages: 18 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-12; Primary Completion 2012-01-11 (Actual); Study Completion 2013-12-05 (Actual)

PRIMARY OUTCOMES:
Incidence of major adverse cardiac event (MACE) (MACE defined as: cardiac death, cardiac arrest, myocardial infarction, sustained ventricular arrhythmias, pulmonary edema, acute heart failure, unstable angina and major bleeding) | Outcome measures will generally be assessed at Baseline, Month 3, Month 6 and Month 12

SECONDARY OUTCOMES:
Left ventricular ejection fraction (LVEF) (As determined by Echo, Cardiac CT and SPECT) | Outcome measures will generally be assessed at Baseline, Month 3, Month 6 and Month 12. CT and SPECT are only assessed at Baseline and Month 6.
Change in LV and RV dimensions and in LV volumes (As determined by Echo, Cardiac CT and SPECT) | Outcome measures will generally be assessed at Baseline, Month 3, Month 6 and Month 12. CT and SPECT are only assessed at Baseline and Month 6.
Wall Motion Score Index (WMSI) (As determined by Echo, Cardiac CT and SPECT) | Outcome measures will generally be assessed at Baseline, Month 3, Month 6 and Month 12. CT and SPECT are only assessed at Baseline and Month 6.
Assessment of myocardial perfusion in ischemic patient cohort, only (As determined by SPECT) | Baseline and Month 3
Exercise tolerance (6 minute walk test) | Outcome measures will generally be assessed at Baseline, Month 3, Month 6 and Month 12
Heart failure status (As determined by New York Heart Association (NYHA) heart failure status (NYHA) class and Brain Natriuretic Peptide [BNP]) | Outcome measures will generally be assessed at Baseline, Month 3, Month 6 and Month 12
Angina status (As determined by Canadian Cardiovascular Society (CCS) classification and Troponin I Levels) | Outcome measures will generally be assessed at Baseline, Month 3, Month 6 and Month 12
Quality of life (As determined by Minnesota Living with Heart Failure Questionnaire [MLHFQ]) | Outcome measures will generally be assessed at Baseline, Month 3, Month 6 and Month 12
Pulmonary function (As determined by metabolic stress test) | Baseline, Month 6 and Month 12
Device implantation, transplantation and positive inotrope use (As determined by incidence rates) | Outcome measures will generally be assessed at Baseline, Month 3, Month 6 and Month 12
AICD firing rate | Outcome measures will generally be assessed at Baseline, Month 3, Month 6 and Month 12
Changes in medication for heart failure | Outcome measures will generally be assessed at Baseline, Month 3, Month 6 and Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Henry, MD, Principal Investigator — Minneapolis Heart Institute Foundation
Locations (3):
- United States (3):
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - University Hospitals, Case Western Reserve University, Cleveland, Ohio
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Derived] Henry TD, Traverse JH, Hammon BL, East CA, Bruckner B, Remmers AE, Recker D, Bull DA, Patel AN. Safety and efficacy of ixmyelocel-T: an expanded, autologous multi-cellular therapy, in dilated cardiomyopathy. Circ Res. 2014 Sep 26;115(8):730-7. doi: 10.1161/CIRCRESAHA.115.304554. Epub 2014 Aug 20. PMID 25142002